CLINICAL TRIAL: NCT06908343
Title: The Associations Between Psychotherapy Expectations and Distress Among Adults Hospitalized in Psychiatric Departments or Treated in the Ambulatory/Community Clinics and Their Therapists.
Brief Title: Psychotherapy Expectations and Distress Among Mental Health Patients and Their Therapists.
Status: Recruiting | Type: Observational
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Yuval Bloch, Prof Dana Tzur Bitan, Shalvata Mental Health Center
Other Study IDs: 0012-22 SHA
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Expectancy; Distress, Psychological
Keywords: process expectations; distress; hospitalized patients; psychotherapy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients at Shalvata Mental Health Center

SUMMARY:
Patients will be recruited from the units of Shalvata MHC: closed and open hospitalization unit, and ambulatory units of Shalvata MHC community clinic. Their therapists will be recruited as well. There will be 4 timepoints measurement: baseline, second week, fourth week and after eight weeks (or discharge). Patients will be addressed through the therapeutic staff and the research team will contact them after a conceptually agreement to participate. A member of the research staff will schedule a meeting explaining the research thoroughly and ask the patient/therapist to sign an informed consent. After signing an informed consent, patients will complete several questionnaires at several time points, whereas their therapists will complete measures as well. All scales will be filled using the Qualtrics platform. In hospitalization unit questionnaires will be filled with the aid of the research coordinator, and in the facilities of Shalvata MHC, in face-to-face interaction. During the face-to-face interaction, in case the patient will report suicidal thoughts or plan to a member of the research staff, the therapeutic staff will be notified immediately. patients at community clinics will fill the first measurement in face-to-face interaction and the rest of the questionnaires independently recieveg a link to their mobile phone.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew mother tongue speakers
* Being treated at Shalvata MHC.

Exclusion Criteria:

* Inability to read or comprehend Hebrew due to any reason.
* Agitative patients
* Acute suicidal patients
* Patients in unstable psychotic state

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sample will be comprised of adults hospitalized in psychiatric departments or treated in the ambulatory/community clinics of Shalvata MHC and their therapists.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom Checklist (SCL-10R) | From enrollment, 2 weeks, 4 weeks and 8 weeks after enrolment
  The scale is a shorter version of the SCL-90 , a self-report inventory consist of 90 items that measure psychosomatic and psychological symptoms for the recent week. The shorter version includes 10 items and has been used in several studies for global psychological distress. Participants are asked to rate each item on a 5-point Likert scale (0 = "no at all" to 4 = "extremely") (e.g. feeling blue). Higher score represents more psychopathology. Cronbach's alpha of the scale was 0.87. In the current study we will translate the questionnaire to Hebrew using back-translation.
The Expectations of Active Processes in Psychotherapy Scale (EAPPS) | At enrollment and 8 weeks after enrolment
  The EAPPS is a scale designed to assess expectations about the active processes assumed to facilitates change in psychotherapy. It includes 32 items representing 7 factors: establishment of positive therapist-client relations, verbal processing of therapist-client relations, exploration of unexpressed contents, the ability to share sensitive contents openly and secretly, working through specific emotional problems, therapy fosters resilience and therapy provides tools for cognitive control. Each respondent will be asked to rate their level of agreement with each item as a mechanism therapy work through on a 7-point Likert scale ranging from 1 (Not at all) to 7 (To a large extent). The score for each factor is calculated by the sum of its items. The EAPPS have been developed in Hebrew and translated into English. Cronbach's alpha of the subscales ranged between .66-.85, and internal and external validity has been established.
Outcome expectations (an item from Credibility/Expectancy Questionnaire (CEQ) | From enrollment, 2 weeks, 4 weeks and 8 weeks after enrollment
  for measuring outcome expectations we will use this 6 items scale divided to two parts. The first one addresses what the subject thinks and includes three credibility items rated on a 9-point Likert-type scale. the minimum value is 1 (not at all sure/think the therapy will be useful) and the maximum value is 9 (very useful). Also, one outcome expectancy item rated from 0 to 100% in 10 jumps (e.g. 0, 10%, 20%...).''By the end of the therapy period, how much improvement in your presenting concerns/problems do you think will occur?''. The second part includes two items rated on a 9-point Likert-type scale that addresses to what the subject feels (e.g." By the end of the therapy period, how much improvement in your presenting concerns/problems do you feel will occur?'. For reliability measure, the total scale standardized alpha was r=0.85. This measure was used in several studies for outcome expectations and was correlated with other outcome expectations measures.
The Clinical Global Impressions Scale (CGI). | From enrollment, 2 weeks, 4 weeks and 8 weeks after enrollment
  The scale is being used for clinicians, who are not necessarily researchers, in order to track patient's progress and treatment response over time. It includes two questions: (1) CGI-Severity and (2) CGI-Improvement. The severity question is: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?". Rated on a seven-point scale from 1=normal, not at all ill, to 7=among the most extremely ill patients. The improvement question is: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment." It is important to note there are guidelines for its use.

SECONDARY OUTCOMES:
The Multitheoretical List of Therapeutic Interventions (MULTI). | 2 weeks and 4 weeks after enrollment
  The MULTI is a 30 items questionnaire focused on interventions from eight different psychotherapy orientations (behavioral, cognitive, dialectical behavioral, interpersonal, person centered, psychodynamic, process- experiential, and common factors). Items are rated from 1(not typical at all) to 5 (extremely typical).
The Stanford Expectations of Treatment Scale (SETS) | At enrollment and 6 weeks after enrollment
  assesses positive and negative treatment expectations with 3 items each on 7-point Likert-scales from 0 'Strongly Disagree׳ l' to 6 'Strongly agree'. An example item of positive treatment expectation is "This treatment will be completely effective" and an example of negative treatment expectation is "I have fears about this treatment". The scale demonstrated good reliability (above .81 for both subscales) and predicted a significant amount of outcome variance (between 12% and 18%). The scale will be translated to Hebrew using back translation. For the therapists the word "my" will be replaced by the word "my patient".
Existential Isolation Scale (EIS) | At enrollment and 8 weeks after enrollment
  The EIS measures social isolation resulting from feeling like no one understands you or reacts to the world differently. The scale has 6 items in which the respondent is asked to rate on a 10-point Likert scale, ranging from 0 (strongly disagree) to 9 (strongly agree) (e.g. People do not often share my perspective). The scale test-retest reliability in the validation article was r(144) = .78.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental Health Center, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Younger J, Gandhi V, Hubbard E, Mackey S. Development of the Stanford Expectations of Treatment Scale (SETS): a tool for measuring patient outcome expectancy in clinical trials. Clin Trials. 2012 Dec;9(6):767-76. doi: 10.1177/1740774512465064. Epub 2012 Nov 20. PMID 23169874
- [Background] McCarthy KS, Barber JP. The Multitheoretical List of Therapeutic Interventions (MULTI): initial report. Psychother Res. 2009 Jan;19(1):96-113. doi: 10.1080/10503300802524343. PMID 19065285
- [Background] Pinel, E. C., Long, A. E., Murdoch, E. Q., & Helm, P. (2017). A prisoner of one's own mind: Identifying and understanding existential isolation. Personality and Individual Differences, 105, 54-63.
- [Background] Solomonov N, McCarthy KS, Gorman BS, Barber JP. The Multitheoretical List of Therapeutic Interventions - 30 items (MULTI-30). Psychother Res. 2019 Jul;29(5):565-580. doi: 10.1080/10503307.2017.1422216. Epub 2018 Jan 16. PMID 29336228
- [Background] Rosen CS, Drescher KD, Moos RH, Finney JW, Murphy RT, Gusman F. Six- and ten-item indexes of psychological distress based on the Symptom Checklist-90. Assessment. 2000 Jun;7(2):103-11. doi: 10.1177/107319110000700201. PMID 10868247
- [Background] Derogatis LR, Lipman RS, Covi L. SCL-90: an outpatient psychiatric rating scale--preliminary report. Psychopharmacol Bull. 1973 Jan;9(1):13-28. No abstract available. PMID 4682398
- [Background] Coyne AE, Constantino MJ, Boswell JF, Gaines AN, Kraus DR. Therapist-Level Moderators of Patient-Therapist Match Effectiveness in Community Psychotherapy. Adm Policy Ment Health. 2024 Sep;51(5):738-752. doi: 10.1007/s10488-024-01360-8. Epub 2024 Apr 2. PMID 38565810
- [Background] Constantino MJ, Coyne AE, McVicar EL, Ametrano RM. The relative association between individual difference variables and general psychotherapy outcome expectation in socially anxious individuals. Psychother Res. 2017 Sep;27(5):583-594. doi: 10.1080/10503307.2016.1138336. Epub 2016 Feb 11. PMID 26866269
- [Background] Tzur Bitan D, Lazar A, Siton B. Development of a scale quantifying expectations regarding active processes in therapy: The Expectations of Active Processes in Psychotherapy Scale (EAPPS). Psychiatry Res. 2018 Sep;267:131-139. doi: 10.1016/j.psychres.2018.05.040. Epub 2018 May 21. PMID 29890376
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Guy W. Hamilton Depression Scale. In: ECDEU Assessment Manual for Psychopharmacology. 1976:179-192. Revised 1976, DHEW Publication No. (ADM) 76-338.
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Brugnera A, Constantino MJ, Grossman-Giron A, Ben David T, Tzur Bitan D. Patient and therapist change process expectations: Independent and dyadic associations with psychotherapy outcomes. Psychother Res. 2025 Apr;35(4):627-636. doi: 10.1080/10503307.2024.2328302. Epub 2024 Mar 14. PMID 38484281
- [Background] Tzur Bitan D, Ben David T, Moshe-Cohen R, Kivity Y. Patient-therapist congruence and incongruence of process expectations during psychotherapy. Psychotherapy (Chic). 2021 Dec;58(4):493-498. doi: 10.1037/pst0000410. PMID 34881924
- [Background] Constantino MJ, Boswell JF, Coyne AE, Swales TP, Kraus DR. Effect of Matching Therapists to Patients vs Assignment as Usual on Adult Psychotherapy Outcomes: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Sep 1;78(9):960-969. doi: 10.1001/jamapsychiatry.2021.1221. PMID 34106240
- [Background] Constantino MJ, Aviram A, Coyne AE, Newkirk K, Greenberg RP, Westra HA, Antony MM. Dyadic, longitudinal associations among outcome expectation and alliance, and their indirect effects on patient outcome. J Couns Psychol. 2020 Jan;67(1):40-50. doi: 10.1037/cou0000364. Epub 2019 Jun 17. PMID 31204836